CLINICAL TRIAL: NCT01433874
Title: Maneuvers to Decrease Upper and Shoulder Pain After Gynecologic Laparoscopic Surgery
Brief Title: Decreasing Upper and Shoulder Pain After Laparoscopic Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Yi-Jen, Chen, M.D., Ph D., Department of Obstetrics and Gynecology, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100-03-001
Record Dates: First submitted 2011-06-14; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-07

CONDITIONS: Shoulder Pain; Nausea
Keywords: Shoulder pain; Upper abdominal pain; Laparoscopic surgery; Abdominal fullness
MeSH Terms: conditions — Shoulder Pain; Nausea; Abdominal Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pulmonary recruitment maneuver (Experimental): A pulmonary recruitment maneuver consisting five manual pulmonary inflations was performed with a maximum pressure of 60 cmH2O. The anesthesiologist held the fifth positive pressure inflation for approximately 5 seconds.
  Interventions: Procedure: Pulmonary recruitment maneuver
- Intraperitoneal normal saline infusion (Experimental): The upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500cc we will leave the fluid in the abdominal cavity.
  Interventions: Procedure: Intraperitoneal normal saline infusion
- combined group (Experimental): The upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500cc. Later, a pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure of 60 cmH20. The anesthesiologist held the fifth positive pressure inflation for approximately 5 seconds.
  Interventions: Procedure: combined group
- Control group (Placebo Comparator): Co2 was removed by passive exsufflation through the port site
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Pulmonary recruitment maneuver — A pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure of 60 cmH2O. The anesthesiologist held the fifth positive pressure inflation for approximately 5 seconds.
  Arms: Pulmonary recruitment maneuver
Procedure: Intraperitoneal normal saline infusion — The upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500cc. We will leave the fluid in the abdominal cavity
  Arms: Intraperitoneal normal saline infusion
Procedure: combined group — The upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500cc. Later, a pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure oof 60 cmH2O.
  Arms: combined group
Procedure: Control group — Co2 was removed by passive exsufflation through the port site.
  Arms: Control group

SUMMARY:
Laparoscopic surgery is becoming a major procedure, owing to smaller incisions, shorter hospitalizations, and less post-operative pain as compared with traditional laparotomies. However, there is marked interindividual variability of post-operative shoulder-tip pain following laparoscopic surgery. The incidence of shoulder pain varies from 35% to 80% and ranges from mild to severe. In some cases, it has been reported to last more than 72 hours after surgery.

The hypothesis of post-operative shoulder-tip pain is that carbon dioxide induced phrenic nerve irritation causes referred pain to C4. Therefore, the investigators should try to do is that if the investigators could reduce carbon dioxide retention in the pelvic cavity.

This clinical controlled trial is tried to find out the practical and clinical maneuver to reduce post-operative should-tip pain following laparoscopic surgery.

DETAILED DESCRIPTION:
This clinical controlled trial is tried to find out the practical and clinical maneuver to reduce post-operative upper abdominal and shoulder pain after laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients receive benign gynecological laparoscopic surgery
* American Society of Anesthesiologists(ASA) physical status of patient classification I-II.

Exclusion Criteria:

* The procedure will be required to conversion to laparotomy
* Any cardio-vascular diseases

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The severity and frequency of upper abdominal and shoulder pain after laparoscopic surgery | The first 48 hours after the surgery
  The investigators will follow the patient in the first 48 hours after the surgery. The primary outcome measure of this trial is the severity and frequency of shoulder and upper abdominal pain after laparoscopic surgery.

SECONDARY OUTCOMES:
nausea or abdominal fullness after laparoscopic surgery | The first 38 hours after the surgery
  postoperative illness, such as nausea, vomiting, or abdominal fullness were also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Wen Tsai, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan; Yi-Jen Chen, M.D., Ph D., Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749
- [Result] Esmat ME, Elsebae MM, Nasr MM, Elsebaie SB. Combined low pressure pneumoperitoneum and intraperitoneal infusion of normal saline for reducing shoulder tip pain following laparoscopic cholecystectomy. World J Surg. 2006 Nov;30(11):1969-73. doi: 10.1007/s00268-005-0752-z. PMID 17043939
- [Derived] Tsai HW, Wang PH, Yen MS, Chao KC, Hsu TF, Chen YJ. Prevention of postlaparoscopic shoulder and upper abdominal pain: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):526-531. doi: 10.1097/AOG.0b013e318283fcca. PMID 23635614